CLINICAL TRIAL: NCT00930917
Title: Heat Loss Prevention in Delivery Room: a Prospective, Randomised, Controlled Trial of Polyethylene Caps in Very Preterm Infants
Brief Title: Heat Loss Prevention in Delivery Room Using a Polyethylene Cap
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Daniele Trevisanuto, Azienda Ospedaliera of Padua
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NIDA8
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Hypothermia, Preterm Infants
Keywords: delivery room, polyethylene cap, preterm infant, temperature
MeSH Terms: conditions — Hypothermia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- cap (Experimental): In the cap group, the head of the infant was covered with a polyethylene cap immediately after birth
  Interventions: Device: Polyethylene cap
- wrap (Active Comparator): Infants in the wrap group were placed into the polyethylene bag, while still wet, up to their necks; only the head was dried.
  Interventions: Device: Polyethylene wrap
- conventional group (Other): Infants in the control group were dried completely, according to International Guidelines for Neonatal Resuscitation.
  Interventions: Other: conventional treatment

INTERVENTIONS:
Device: Polyethylene cap — In the cap group, the head of the infant was covered with a polyethylene cap immediately after birth
  Arms: cap
Device: Polyethylene wrap — Infants in the wrap group were placed into the polyethylene bag, while still wet, up to their necks; only the head was dried.
  Arms: wrap
Other: conventional treatment — Infants in the control group were dried completely, according to International Guidelines for Neonatal Resuscitation.
  Arms: conventional group

SUMMARY:
It is apparent that the head of a preterm infant should not be left uncovered, however it remains unclear whether covering the head of a preterm baby with plastic wrapping is effective in preventing heat loss.

We conducted a prospective, randomised, controlled trial in very preterm infants to evaluate if a polyethylene cap prevents heat loss after delivery better than polyethylene occlusive wrapping and conventional drying. Furthermore, we assessed body temperature 1 hour after admission to Neonatal Intensive Care Unit (NICU) to evaluate whether the polyethylene cap prevents postnatal heat loss.

DETAILED DESCRIPTION:
The primary outcome measure was axillary temperature taken on admission to the NICU (immediately after cap and wrap removal) and again 1 hour later. Axillary temperature was measured using a digital thermometer (Terumo Digital Clinical Thermometer C202, Terumo Corporation, Tokio, Japan). The occurrence of hypothermia, defined as axillary temperature less then 36.4°C, on NICU admission was also evaluated.

Secondary outcomes included mortality prior to hospital discharge, presence of major brain injury (sonographic evidence of intraventricular hemorrhage with ventricular dilatation, parenchymal hemorrhagic infarction, or periventricular leukomalacia), tracheal intubation at birth, Apgar scores, delivery to admission time, blood gas analysis and serum glucose concentration on NICU admission.

ELIGIBILITY:
Inclusion Criteria:

* infants <29 weeks' gestation born in the study center.

Exclusion Criteria:

* congenital anomalies with open lesions (e.g. gastroschisis, meningomyelocele) and babies whose delivery was not attended by the neonatal team.

Ages: 1 Minute to 3 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Axillary temperature taken on admission to the NICU (immediately after cap and wrap removal) and again 1 hour later. | Admission to the NICU

SECONDARY OUTCOMES:
Mortality prior to hospital discharge, presence of major brain injury, tracheal intubation at birth, Apgar scores, delivery to admission time, blood gas analysis and serum glucose concentration on NICU admission. | NICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Trevisanuto, MD, Principal Investigator — Azienda Ospedaliera of Padua

REFERENCES:
- [Derived] Trevisanuto D, Doglioni N, Cavallin F, Parotto M, Micaglio M, Zanardo V. Heat loss prevention in very preterm infants in delivery rooms: a prospective, randomized, controlled trial of polyethylene caps. J Pediatr. 2010 Jun;156(6):914-917.e1. doi: 10.1016/j.jpeds.2009.12.021. Epub 2010 Mar 15. PMID 20227728